CLINICAL TRIAL: NCT06039202
Title: A Phase 2, Randomized, Open Label Study to Evaluate Efficacy, Safety, and Tolerability of CA102N Combined With Trifluridine/Tipiracil (TAS-102) Compared to Bevacizumab Combined With TAS-102 in Subjects With Metastatic Colorectal Cancer (mCRC) Who Failed the Standard Treatment
Brief Title: Phase 2 Study of CA102N Combined With TAS-102 Compared to Bevacizumab Combined With TAS-102 in Subjects With Relapsed and/or Refractory Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Holy Stone Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-CA102N-103
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Up to 100 subjects will be enrolled in this study (including drop-out subjects), with 50 subjects assigned to each treatment arm.
  For arm 1, subjects will receive the assigned dose level of CA102N in combination with trifluridine/tipiracil (TAS-102). For Arm 2, subjects will receive bevacizumab in combination with trifluridine/tipiracil (TAS-102)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CA102N plus Trifluridine/tipiracil (TAS-102) (Experimental): CA102N administered as 0.72 mg/kg of nimesulide equivalents on Days 1 and 15 of each 28-day cycle in combination with TAS-102 at 35 mg/m2/dose orally twice daily (BID) on Days 1 through 5 and Days 8 through 12 of each 28-day cycle. Administration sequence will be CA102N then TAS-102 (IV then oral)
  Interventions: Drug: CA102N; Drug: TAS-102
- Bevacizumab plus Trifluridine/tipiracil (TAS-102) (Active Comparator): bevacizumab 5 mg/kg on Days 1 and 15 of each 28-day cycle in combination with 35 mg/m2 of TAS-102 orally twice daily (BID) on Days 1 through 5 and Days 8 through 12 of each 28-day cycle. Administration sequence will be bevacizumab then TAS-102 (IV then oral)
  Interventions: Drug: TAS-102; Biological: Bevacizumab

INTERVENTIONS:
Drug: CA102N — CA102N is a covalently bound conjugate of the biological polymer sodium hyaluronate (NaHA) and nimesulide (Nim)
  Other Names: Nim-HA cinjugate
  Arms: CA102N plus Trifluridine/tipiracil (TAS-102)
Drug: TAS-102 — TAS-102 is a cytotoxic combination treatment of 2 drugs: trifluridine, a thymidine-based nucleoside analogue, and tipiracil an inhibitor of thymidine phosphorylase.
  Other Names: Trifluridine/tipiracil
Biological: Bevacizumab — Bevacizumab recombinant humanized monoclonal antibody that binds and neutralizes circulating vascular endothelial growth factor (VEGF)-A.
  Arms: Bevacizumab plus Trifluridine/tipiracil (TAS-102)

SUMMARY:
HS-CA102N-103 is a Phase 2, randomized, open label study to evaluate efficacy, safety, and tolerability of CA102N combined with trifluridine/tipiracil (TAS-102) compared to bevacizumab combined with TAS-102 in subjects with metastatic colorectal cancer (mCRC) who failed the standard treatment (for eg, cancer that has relapsed after or is refractory to fluoropyrimidine, oxaliplatin and irinotecan-based chemotherapy).

DETAILED DESCRIPTION:
HS-CA102N-103 is a Phase 2, randomized, open label study to evaluate efficacy, safety, and tolerability of CA102N combined with trifluridine/tipiracil (TAS-102) compared to bevacizumab combined with TAS-102 in subjects with metastatic colorectal cancer (mCRC) who failed the standard treatment (for eg, cancer that has relapsed after or is refractory to fluoropyrimidine, oxaliplatin and irinotecan-based chemotherapy).

In this study, the safety, tolerability, and PFS of CA102N in combination with TAS-102 compared to bevacizumab combined with TAS-102 will be evaluated in up to 100 subjects with metastatic colorectal cancer who have previously received fluoropyrimidine, oxaliplatin, and irinotecan-based chemotherapy, an anti-vascular endothelial growth factor (VEGF) biological therapy, and if RAS wild-type mCRC, an anti-epidermal growth factor receptor (EGFR) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥20 years in Taiwan, and Korea, or those aged ≥18 years in the US, at the time the ICFs are signed. (Please follow local regulatory requirements if the legal age of consent for study participation is different).
* Have relapsed after, intolerant to, or are refractory to fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and if RAS wild-type, an anti-EGFR therapy.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Presence of at least one measurable lesion (minimum 10 mm) assessed by the Investigator per RECIST version 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions after the end of radiotherapy.
* Has a life expectancy of ≥3 months.
* Women of childbearing potential and men with partners of childbearing potential must agree to use a highly effective means of contraception from study entry through at least 6 months after the last dose of CA102N.

Exclusion Criteria:

* History of hypersensitivity or hepatotoxic reactions to nimesulide or to any excipient.
* History or presence of a bleeding tendency or disorder.
* History of gastrointestinal bleed or perforation related to previous nonsteroidal anti-inflammatory drugs (NSAIDs) or bevacizumab.
* Presence or history of recurrent peptic ulcer or hemorrhage (2 or more distinct episodes of proven ulceration or bleeding).
* History of cerebrovascular or other active bleeding.
* Myocardial infarction within the last 12 months prior to the first dose of study drug, severe/unstable angina, symptomatic congestive heart failure New York Heart Association Class III or IV.
* History of a serious cardiac arrhythmia requiring treatment. Subjects whose arrhythmia is well-controlled (eg, by ablation or medical therapy) may be considered for enrollment after discussion with the study medical monitor.
* Has had clinically significant lung disease (eg, interstitial pneumonia, interstitial lung disease, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) requiring continuous systemic corticosteroid treatment for 6 months before Screening or who are suspected to have such diseases by imaging at Screening.
* Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks prior to Screening, or subject who continues to have a peritoneal/pleural/pericardial drainage catheter post-surgery at the time of informed consent signature.
* History of allogeneic transplantation requiring immunosuppressive therapy.
* Presence of uncontrolled infections.
* Known positive test for hepatitis B, hepatitis C or human immunodeficiency virus. Testing is not required for protocol eligibility. Subjects who have received curative therapy for HCV with no detectable viral load are not excluded.
* Has clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids and stable brain metastases at least 3 months may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
* Pregnant or breast feeding or intends to become pregnant during the study.
* Unresolved toxicity of greater than or equal to NCI-CTCAE (version 5.0) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced peripheral neurotoxicity).
* Has a concomitant medical condition that would increase the risk of toxicity or confine the interpretation of efficacy or safety in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of CA102N in combination with trifluridine/tipiracil (TAS-102) by progression free survival (PFS) rate. | 16 weeks after first treatment.
Number of subjects with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | one year after first treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 16 weeks after first treatment.
  To evaluate the efficacy of CA102N in combination with trifluridine/tipiracil (TAS-102) by disease control rate.
Overall response rate (ORR) | 16 weeks after first treatment.
  To evaluate the efficacy of CA102N in combination with trifluridine/tipiracil (TAS-102) by overall response rate.
Maximum Plasma Concentration [Cmax] of CA102N when used in combination with trifluridine/tipiracil (TAS-102) | 16 weeks after first treatment.
To evaluate the efficacy of CA102N in combination with trifluridine/tipiracil (TAS-102) by overall survival (OS). | one year after first treatment.

OTHER OUTCOMES:
Protein expression level of pharmacodynamic biomarkers | 16 weeks after first treatment.
Quality of life measured by European Organization for the research and treatment of cancer quality of life questionnaire (EORTC QLQ-C30). | one year after first treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pant S, Dragovich T, Lieu C, Jimeno A, Kundranda M, Menter D, Tchaparian E, Chen YC, Kopetz S. Phase 1 study of the safety, pharmacokinetics, and preliminary efficacy of CA102N as monotherapy and in combination with trifluridine-tipiracil in patients with locally advanced or metastatic solid tumors. Invest New Drugs. 2023 Feb;41(1):25-34. doi: 10.1007/s10637-022-01308-5. Epub 2022 Nov 4. PMID 36331676
- See also: The result of phase I study — https://pubmed.ncbi.nlm.nih.gov/36331676/